CLINICAL TRIAL: NCT05544942
Title: GCWB1001 12 Weeks, Multi -Tube, Randomized Assignment, Double -Eye, Placebo Control Human Application Test for Evaluating the Effectiveness and Safety of the Respiratory Health Health
Brief Title: GCWB1001 Evaluates the Effectiveness and Safety of Respiratory Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Wellbeing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GCWB109
Record Dates: First submitted 2022-09-05; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Respiratory Symptoms
MeSH Terms: conditions — Signs and Symptoms, Respiratory | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GCWB1001 (Experimental): 1 capsule once a day
  Interventions: Dietary Supplement: Lactobacillus plantarum
- Placebo (Active Comparator): 1 capsule once a day
  Interventions: Other: maltodextrin

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum — 1 capsule once a day
  Arms: GCWB1001
Other: maltodextrin — 1 capsule once a day
  Arms: Placebo

SUMMARY:
This human application test was designed to evaluate the effectiveness and safety of the losing suction tendon, compared to the control food when the GCWB1001 was consistent with the symptoms of the respiratory symptoms of mildness.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of screening, 19 or 70 years
2. Those who have two or more symptoms of cough, sputum, lake striking or chest stuffy for more than one month, and BCSS at 3 or more
3. Those with FEV 1 /FVC 70 or higher
4. Those who agreed to participation in this human application test before the beginning of the human test and signed in the Informed Consent Form

Exclusion Criteria:

1. Severe cardiovascular, immune system, gastrointestinal and biliary meters, kidney and urinary systems, Those who are currently treated with neurological system, musculoskeletal system, mental, infectious diseases and malignant tumors
2. Those who have clinically significant respiratory diseases findings as a result of chest X-ray shooting
3. Those who have been diagnosed with chronic obstructive pulmonary disease (COPD) or asthma
4. Chronic bronchitis (BCSS 9 or more points or more Those who have continuous cough, sputum symptoms for more than 3 months)
5. A person who has a respiratory symptom due to virus or bacteria within 4 weeks of visit (Influenza, Corona Virus infection 19, pneumonia, acute infection, etc.) However, if the corona virus infection 19 has worsened or new symptoms of respiratory symptoms occur (However, if there are no additional respiratory symptoms caused by corona-19 infections, you can participate after 4 weeks after isolation. In the case of additional respiratory symptoms, the symptoms improve and can be participated if they have been restored to the time of recovery so that there is no difference compared to before infection.)
6. Those who take drugs for the purpose of taking immunosuppressive agents, or for the purpose of regulating Jinhae expectoration within 4 weeks of visit.
7. Those who take health functional foods related to improvement of respiratory health within 2 weeks of visit 1
8. Those who administered antibiotics within 2 weeks of visiting 1
9. Probiotics and those who consistently consume lactic acid bacteria products (4 or more times a week) within 2 weeks
10. Those who are less than 6 months after smokers or smoking cessation
11. Less than 4 weeks of visit, a person who falls under alcohol with an average of 30 g (210 shares) per day (210 weeks), an average of 20 g or more (140 shares) per day (140 shares)
12. Those who are more than twice the summit of Creatinine.
13. AST (G OT) or ALT (GPT) is three times more than the normal upper limit of the embodiment
14. Inconsidable high blood pressure patients systolic blood pressure 160 mmHg or higher or relaxation blood pressure 100 mmHg or higher, test target 10 minutes stabilization
15. Ungodined diabetic patient empathy 180 mg/dL or more
16. Those who are pregnant or have a planning plan for lactation or this human application period
17. Those who have been administered to include other arbitral clinical trial applications within 3 months of visitor and have received food for adoption of drugs for clinical trials. Those who plan to participate
18. Those who are sensitive or allergic to food ingredients for this human application
19. Those who judge that the tester is inadequate for other reasons

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change amoust of BCSS | week -2, 6 and 12
  The comparison of the bcss change in the before and after the intake of the BCSS is analyzed using the Paired T-TEST, and the degree of change between the test group and the control group at each point of view is the Two Sample T-Test and the Wilcoxon Rank Sum test It is conducted to evaluate whether there is a significant difference.

SECONDARY OUTCOMES:
Change amoust of Lung function (FVC, FEV1, FEV1/FVC) | week -2, 6 and 12
  The comparison of the Lung function (FVC, FEV1, FEV1/FVC) change in the before and after the intake of the Lung function (FVC, FEV1, FEV1/FVC) is analyzed using the Paired T-TEST, and the degree of change between the test group and the control group at each point of view is the Two Sample T-Test and the Wilcoxon Rank Sum test It is conducted to evaluate whether there is a significant difference.
Change amoust of SGRQ | week -2, 6 and 12
  The comparison of the SGRQ change in the before and after the intake of the SGRQ is analyzed using the Paired T-TEST, and the degree of change between the test group and the control group at each point of view is the Two Sample T-Test and the Wilcoxon Rank Sum test It is conducted to evaluate whether there is a significant difference.
Change amoust of VAS | week -2, 6 and 12
  The comparison of the VAS change in the before and after the intake of the VAS is analyzed using the Paired T-TEST, and the degree of change between the test group and the control group at each point of view is the Two Sample T-Test and the Wilcoxon Rank Sum test It is conducted to evaluate whether there is a significant difference.
Change amoust of blood biomarker (TNF-α, IgE, IL-6, IL-10, IFN-γ) | week -2 and 12
  The comparison of the blood biomarker change in the before and after the intake of the blood biomarker is analyzed using the Paired T-TEST, and the degree of change between the test group and the control group at each point of view is the Two Sample T-Test and the Wilcoxon Rank Sum test It is conducted to evaluate whether there is a significant difference.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - HALLYM UNIV. Chuncheon MEDICAL CENTER, Chuncheon
  - Hallym Univ. Medical Center, Gyeonggi-do
  - Chungbuk national university hospital, Jungbuk
  - Hanyang University Seoul Hospital, Seoul